CLINICAL TRIAL: NCT05255874
Title: The Effect of Aromatherapy Applied to the Patients in the Urodynamic Procedure on Anxiety and Serum Cortisol Levels
Brief Title: The Effect of Aromatherapy Applied to the Patients in the Urodynamic Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Elife Kettas Dolek, Urology Polyclinic Responsible Nurse, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersınUnıver
Record Dates: First submitted 2022-02-14; First posted 2022-02-25 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Anxiety
Keywords: Anxiety; Aromatherapy; Urodynamic; Serum Cortisol
MeSH Terms: conditions — Anxiety Disorders | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy Group (Experimental): Patients in the study group will rest for 5 minutes before and after the urodynamics procedure. All patients will be asked to fill in the 'Spielberger State Anxiety Scale' before and after the urodynamic procedure. Before and after the procedure, blood pressure, heart rate, respiratory rate, peripheral oxygen saturation will be measured. Blood will be drawn for serum cortisol level. In addition to the routine treatment and care practices of the unit, aromatherapy will be applied to the patients included in the study group. Aromatherapy application will be applied to all patients by the same researcher. Aromatherapy application will be started 5 minutes before the urodynamic procedure after the patient is taken to the urodynamic room, and lavender essential oil (3 drops in 300 cc water for 5 cubic meters of room) will be used with a diffuser until the end of the procedure.
  Interventions: Other: Aromatherapy
- Standard of care (No Intervention): Routine treatment and care interventions will be applied to the patients included in the control group during the procedure. Patients in the control group will rest for 5 minutes before and after the urodynamics procedure. All patients will be asked to fill in the 'Spielberger State Anxiety Scale' before and after the urodynamic procedure. Before and after the procedure, blood pressure, heart rate, respiratory rate, peripheral oxygen saturation will be measured. Blood will be drawn for serum cortisol level.

INTERVENTIONS:
Other: Aromatherapy — Patients in the study group will rest for 5 minutes before and after the urodynamics procedure. All patients will be asked to fill in the 'Spielberger State Anxiety Scale' before and after the urodynamic procedure. Before and after the procedure, blood pressure, heart rate, respiratory rate, peripheral oxygen saturation will be measured. Blood will be drawn for serum cortisol level. In addition to the routine treatment and care practices of the unit, aromatherapy will be applied to the patients included in the study group. Aromatherapy application will be applied to all patients by the same researcher. Aromatherapy application will be started 5 minutes before the urodynamic procedure after the patient is taken to the urodynamic room, and lavender essential oil (3 drops in 300 cc water for 5 cubic meters of room) will be used with a diffuser until the end of the procedure.
  Arms: Aromatherapy Group

SUMMARY:
This randomized controlled study is planned to determine the effect of aromatherapy applied to patients in the urodynamic procedure on patients' anxiety and serum cortisol levels.

This study assumes that lavender inhalation in aromatherapy has positive effects on physiological parameters such as blood pressure, heart rate, respiratory rate, serum cortisol level, as well as reducing stress and anxiety.

DETAILED DESCRIPTION:
98 patients in each group will be included in the study (Aromatherapy group=49; Control group=49). In addition to the routine treatment and care practices of the unit, aromatherapy will be applied to the patients included in the study group. Aromatherapy application will be applied to all patients by the same researcher. Aromatherapy application will be started 5 minutes before the urodynamic procedure after the patient is taken to the urodynamics room and lavender essential oil will be used with a diffuser until the end of the procedure. Routine treatment and care interventions will be applied to the patients included in the control group during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Those who signed the 'Informed Voluntary Consent Form' to participate in the research,
* 18 years and older,
* Conscious, oriented and cooperative,
* Able to communicate
* Urodynamic procedure applied,
* No problem in sense of smell,
* No chronic respiratory disease (lung cancer, chronic obstructive pulmonary disease, asthma, chronic bronchitis, etc.),
* No history of dermatitis against cosmetic odor,
* Patients without a known history of allergy to the essential oil used

Exclusion Criteria:

* Those who did not sign the "Informed Consent Form" to participate in the research,
* Under 18 years of age,
* Unconscious, without orientation and cooperation,
* Unable to communicate,
* Urodynamic procedure is not applied.
* Having problems with the sense of smell,
* Having chronic respiratory disease (lung cancer, chronic obstructive pulmonary disease, asthma, chronic bronchitis, etc.),
* Having a history of dermatitis against cosmetic odor,
* Having a trait anxiety scale score of 60 and above,
* Patients with a known history of allergy to the essential oil used

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Anxiety evaluated using the State Anxiety Scale | Change from Baseline (before implementation) and within 5 minutes after procedure
  Scores ranging from 20 to 80 points are obtained in the scale. In the total score obtained from the scale in scoring the scale, 0-19 points indicate the absence of anxiety, 20-39 points indicate mild anxiety, 40-59 points indicate moderate anxiety, and 60-79 points indicate severe anxiety level. Higher state anxiety scores indicate that anxiety level is also high

SECONDARY OUTCOMES:
Change systolic and diastolic blood pressure | Change from Baseline (before implementation) and within 5 minutes after procedure
  Before and after the procedure systolic and diastolic blood pressure will be measured.
Change heart rate | Change from Baseline (before implementation) and within 5 minutes after procedure
  Before and after the procedure heart rate will be measured.
Change respiratory rate | Change from Baseline (before implementation) and within 5 minutes after procedure
  Before and after the procedure respiratory rate will be measured.
Change peripheral oxygen saturation | Change from Baseline (before implementation) and within 5 minutes after procedure
  Before and after the procedure peripheral oxygen saturation will be measured.
Change serum cortisol level | Change from Baseline (before implementation) and within 5 minutes after procedure
  Before and after the procedure blood will be drawn for serum cortisol level.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLAY ALTUN UĞRAŞ, Study Director — MERSİN UNIVERSITY
Locations (1):
- Elife Kettaş Dölek, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ozel BZ, Quevedo A, Jung C, Shirazi F, Dancz CE. Lavender Aromatherapy for Anxiety and Pain During Multichannel Urodynamics: A Randomized Controlled Pilot Trial. Female Pelvic Med Reconstr Surg. 2021 Nov 1;27(11):654-658. doi: 10.1097/SPV.0000000000001032. PMID 33626029